CLINICAL TRIAL: NCT00677573
Title: Comparison of Urinary Purified Follicle-Stimulating Hormone (FSH) and Rec-FSH Among Poor Responders Undergoing Ovarian Stimulation With GnRH Antagonist
Brief Title: Efficacy of Urinary Follicle-Stimulating Hormone (FSH) Among Poor Responders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: German Hospital, Istanbul (Other)
Collaborators: Bahceci Women Health Care Center (Unknown)
Responsible Party: German Hospital, Istanbul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ughno1
Record Dates: First submitted 2008-05-09; First posted 2008-05-14 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Infertility
Keywords: ART; poor responder; GnRH antagonist; Gonadotropins
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UrFSH (Active Comparator)
  Interventions: Drug: Fostimon

INTERVENTIONS:
Drug: Fostimon — 450 IU for 4 days then adjusted

SUMMARY:
We proposed to compare outcomes in women with DOR undergoing ART with rec-FSH + u-HMH with those with u-FSH only in GnRH antagonist protocols.

ELIGIBILITY:
Inclusion Criteria:

* At least one trial with adequate ovarian stimulation resulted by 4 or less oocytes retrieval.

Exclusion Criteria:

* High responder patients

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2008-05; Primary Completion 2008-10 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate per embryo transfer | 6 months

SECONDARY OUTCOMES:
number of oocytes retrieved | per patient

CONTACTS AND LOCATIONS:
Locations (1):
- Alman Hastanesi, Istanbul, Istanbul, Turkey (Türkiye)